CLINICAL TRIAL: NCT04814277
Title: Accuracy Evaluation for Software-based Visualization of GPi/GPe Anatomical Brain Structure Using Surgical Information Sciences Inc. Algorithms
Brief Title: Accuracy Evaluation of SIS Software-based Visualization of New Anatomical Brain Structure
Status: Completed | Type: Observational
Sponsor: Surgical Information Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DOC-0055
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Software Evaluation for Visualizing Anatomical Structures Not Typically Identified on Clinical MR Images

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- MRI Data Collection: A group of 34 subjects will be scanned on a 3Tesla (3T) and on a 7T MRI scanner. The images will be compared.

SUMMARY:
SIS has developed a software technology, based on machine learning and image processing, designed to enhance standard clinical images for the visualization of anatomical structures.

DETAILED DESCRIPTION:
A cohort of 34 subjects will be scanned on a clinical MRI scanner as well as on a 7 Tesla (7T) scanner. Images acquired on the 7T allow to visualize anatomical structures that are not easily identified on standard clinical images.

SIS software will be used to visualize selected anatomical features on the clinical image and the results will be compared with the images in the same subject obtained from the 7T MRI.

ELIGIBILITY:
Inclusion Criteria:

* All subjects that are willing to be scanned on a 3T and 7T MRI scanners and are not excluded by the exclusion criteria below.

Exclusion Criteria:

1. MRI exclusion criteria for 7T scans: presence of any metallic clip(s) or implantable medical devices (e.g,. heart valve, aneurysm clip, coils or surgery, renal or aortic clips, shunts, stents or stent grafts, metal mesh/coil implants, neurostimulator, insulin pump, IVC filter, artificial knee or hip, metal plates, pins, screws or wires anywhere in the body, any other metal implants, etc.
2. Pregnant women.
3. Subject under the age of 18.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of 34 adults who will be scanned on a 3T and 7T MRI to obtain anatomical images of their brain.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Validation of the accurate visualization of brain structure based on SIS algorithms - 1 | Through study completion, up to 1 year
  Difference in distance between brain structure center of mass (COM)
Validation of the accurate visualization of brain structure based on SIS algorithms - 2 | Through study completion, up to 1 year
  Difference in distance between brain structure mean surface area
Validation of the accurate visualization of brain structure based on SIS algorithms - 3 | Through study completion, up to 1 year
  Difference in Dice Coefficient between measured brain structures

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Information Sciences, Plymouth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No